CLINICAL TRIAL: NCT06608095
Title: A Multicenter, Single-Blind Randomized Controlled Trial of TTM(Target Temperature Management) in Adults With ECPR(Extracorporeal Cardiopulmonary Resuscitation)
Brief Title: Efficacy and Safety of TTM in Adults With ECPR.
Acronym: TTM、ECPR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Qingbian Ma, MD, Director of the Emergency Department, Peking University Third Hospital, Peking University Third Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00006761-M2022581
Record Dates: First submitted 2023-10-20; First posted 2024-09-23 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Cardiac Arrest
Keywords: cardiac arrest; extracorporeal cardiopulmonary resuscitation; hypothermia; normothermia; clinical outcome; randomized controlled trial
MeSH Terms: conditions — Heart Arrest; Hypothermia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hypothermia group (Experimental): Combined target temperature management (TTM) in patients undergoing extracorporeal cardiopulmonary resuscitation (ECPR) and with a target temperature control of 34°C.
  Interventions: Behavioral: hypothermia group
- normothermia group (Experimental): Combined target temperature management (TTM) in patients undergoing extracorporeal cardiopulmonary resuscitation (ECPR) and with a target temperature control of 36.5-37.2°C.
  Interventions: Behavioral: normothermia group

INTERVENTIONS:
Behavioral: hypothermia group — Minimize the temperature of the thermometric tank or thermometric catheter for rapid temperature control. Use a thermometric catheter to monitor changes in the patient's core body temperature in real time. When the core body temperature drops to 34 ℃, adjust the target temperature of the temperature-controlled water tank to 34 ℃ and adjust the target temperature of the temperature-controlled water tank in real time according to the patient's core body temperature. Keep the core body temperature around 34 ℃. Maintain the body temperature at 34℃ for at least 24 hours after the patient resumes autonomous circulation. After the patient has resumed voluntary circulation for 24 hours, the rewarming process can begin. The target temperature of the temperature control tank will increase at a rate of 0.2°C/h. After reaching 36°C, maintain the current temperature. Once 36°C is reached, the current temperature is maintained until autonomic circulation has been restored for 5 days.
  Arms: hypothermia group
Behavioral: normothermia group — Set the temperature of the temperature-controlled water tank or the in vivo cooling catheter to 37°C to maintain the patient's core temperature between 36.5-37.5°C. Real-time monitoring of the patient's core temperature changes through the thermometric urinary catheter, and real-time adjustment of the temperature of the temperature-controlled water tank. The patient's temperature was maintained between 36.5-37.5°C after the patient resumed voluntary circulation until the end of temperature control 5 days after the recovery of voluntary circulation.
  Arms: normothermia group

SUMMARY:
Investigators hypothesize that there is a difference in the 30-day survival rate and good neurological outcome rate between two groups of cardiac arrest patients undergoing ECPR, one group receiving hypothermia and the other group receiving normothermia. Among the patients undergoing extracorporeal cardiopulmonary resuscitation, after screening with inclusion criteria as well as exclusion criteria, informed consent for the experiment was signed and randomly assigned into 2 groups. One group underwent extracorporeal cardiopulmonary resuscitation combined with hypothermia (34°C) and the other group underwent extracorporeal cardiopulmonary resuscitation combined with normothermia (36.5-37.5℃). Information related to the prognosis of the participants in both groups was obtained, evaluated statistically, and final conclusions were drawn.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥18 and ≤60 years;
2. Patients with in-hospital and out-of-hospital cardiac arrest of any initial rhythm;
3. Patients who have received cardiopulmonary resuscitation for >10 minutes without achieving return of spontaneous circulation;
4. Patients with a reversible cause of cardiac arrest (acute myocardial infarction, pulmonary embolism, all initial defibrillatable rhythm, cardiomyopathy);

Exclusion Criteria:

1. cardiac arrest due to trauma;
2. pregnant and lactating women;
3. unwitnessed cardiac arrest;
4. out-of-hospital cardiac arrest not receiving CPR within 5 minutes;
5. > 60 minutes from the onset of cardiac arrest to the initiation of extracorporeal cardiopulmonary resuscitation;
6. achievement of return of spontaneous circulation before the start of external cardiopulmonary resuscitation;
7. intracranial hemorrhage or suspected intracranial hemorrhage;
8. pre-existing neurologic impairment (CPC ≥ 3) prior to the onset of cardiac arrest;
9. those with end-stage heart failure;
10. those with new-onset cerebral hemorrhage or cerebral infarction;
11. other vascular conditions such as severe plaque in bilateral femoral arteries that cause difficulty in tube placement;
12. patients with combined malignant tumors;
13. other serious diseases with a life expectancy of <1 year;
14. refusal to perform extracorporeal cardiopulmonary resuscitation and/or target temperature administrators.
15. Temperature <30°C.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 146 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
30-day survival outcomes | 30 days after randomization
  All-cause survival rate of patients on day 30 after randomization.
30-day neurologic function outcomes | 30 days after randomization
  Rate of patients with good neurological outcome at day 30 of randomization.Good neurological outcome is defined as a cerebral performance category(CPC) score of 1 or 2.

SECONDARY OUTCOMES:
prolong follow-up survival outcome | 90 days and 6 months after randomization
  survival rate
prolong follow-up neurologic outcome | 30 days, 3 months, and 6 months after randomization
  Modified Rankin scale neurologic function scores and cerebral performance category(CPC) scores at 30 days, 3 months, and 6 months after randomization.Modified Rankin scale neurologic function scores assesses the poststroke sequelae, ranges from 0 (no symptoms) to 6 (death), and establishes the patient's functional independence (from 0 to 2) or dependence (from 3 to 5).Cerebral performance category(CPC) scores define a good outcome as a CPC score of 1 or 2, and a poor outcome (severe neurological disability, persistent vegetative state or death) as CPC scores 3, 4, or 5.
Incidence of any bleeding, infection, arrhythmia, acute kidney injury and seizure [Safety and Tolerability] | 30 days after randomization

CONTACTS AND LOCATIONS:
Locations (1):
- Emergency Dept of Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Merchant RM, Topjian AA, Panchal AR, Cheng A, Aziz K, Berg KM, Lavonas EJ, Magid DJ; Adult Basic and Advanced Life Support, Pediatric Basic and Advanced Life Support, Neonatal Life Support, Resuscitation Education Science, and Systems of Care Writing Groups. Part 1: Executive Summary: 2020 American Heart Association Guidelines for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Circulation. 2020 Oct 20;142(16_suppl_2):S337-S357. doi: 10.1161/CIR.0000000000000918. Epub 2020 Oct 21. No abstract available. PMID 33081530
- [Background] Kirkegaard H, Taccone FS, Skrifvars M, Soreide E. Postresuscitation Care after Out-of-hospital Cardiac Arrest: Clinical Update and Focus on Targeted Temperature Management. Anesthesiology. 2019 Jul;131(1):186-208. doi: 10.1097/ALN.0000000000002700. PMID 31021845
- [Background] Nagao K, Nonogi H, Yonemoto N, Gaieski DF, Ito N, Takayama M, Shirai S, Furuya S, Tani S, Kimura T, Saku K; Japanese Circulation Society With Resuscitation Science Study (JCS-ReSS) Group*. Duration of Prehospital Resuscitation Efforts After Out-of-Hospital Cardiac Arrest. Circulation. 2016 Apr 5;133(14):1386-96. doi: 10.1161/CIRCULATIONAHA.115.018788. Epub 2016 Feb 26. PMID 26920493
- [Background] Kennedy JH. The role of assisted circulation in cardiac resuscitation. JAMA. 1966 Aug 22;197(8):615-8. No abstract available. PMID 5953090
- [Background] Panchal AR, Bartos JA, Cabanas JG, Donnino MW, Drennan IR, Hirsch KG, Kudenchuk PJ, Kurz MC, Lavonas EJ, Morley PT, O'Neil BJ, Peberdy MA, Rittenberger JC, Rodriguez AJ, Sawyer KN, Berg KM; Adult Basic and Advanced Life Support Writing Group. Part 3: Adult Basic and Advanced Life Support: 2020 American Heart Association Guidelines for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Circulation. 2020 Oct 20;142(16_suppl_2):S366-S468. doi: 10.1161/CIR.0000000000000916. Epub 2020 Oct 21. No abstract available. PMID 33081529
- [Background] Chen YS, Lin JW, Yu HY, Ko WJ, Jerng JS, Chang WT, Chen WJ, Huang SC, Chi NH, Wang CH, Chen LC, Tsai PR, Wang SS, Hwang JJ, Lin FY. Cardiopulmonary resuscitation with assisted extracorporeal life-support versus conventional cardiopulmonary resuscitation in adults with in-hospital cardiac arrest: an observational study and propensity analysis. Lancet. 2008 Aug 16;372(9638):554-61. doi: 10.1016/S0140-6736(08)60958-7. Epub 2008 Jul 4. PMID 18603291
- [Background] Hypothermia after Cardiac Arrest Study Group. Mild therapeutic hypothermia to improve the neurologic outcome after cardiac arrest. N Engl J Med. 2002 Feb 21;346(8):549-56. doi: 10.1056/NEJMoa012689. PMID 11856793
- [Background] Stub D, Bernard S, Pellegrino V, Smith K, Walker T, Sheldrake J, Hockings L, Shaw J, Duffy SJ, Burrell A, Cameron P, Smit de V, Kaye DM. Refractory cardiac arrest treated with mechanical CPR, hypothermia, ECMO and early reperfusion (the CHEER trial). Resuscitation. 2015 Jan;86:88-94. doi: 10.1016/j.resuscitation.2014.09.010. Epub 2014 Oct 2. PMID 25281189
- [Background] Dankiewicz J, Cronberg T, Lilja G, Jakobsen JC, Levin H, Ullen S, Rylander C, Wise MP, Oddo M, Cariou A, Belohlavek J, Hovdenes J, Saxena M, Kirkegaard H, Young PJ, Pelosi P, Storm C, Taccone FS, Joannidis M, Callaway C, Eastwood GM, Morgan MPG, Nordberg P, Erlinge D, Nichol AD, Chew MS, Hollenberg J, Thomas M, Bewley J, Sweet K, Grejs AM, Christensen S, Haenggi M, Levis A, Lundin A, During J, Schmidbauer S, Keeble TR, Karamasis GV, Schrag C, Faessler E, Smid O, Otahal M, Maggiorini M, Wendel Garcia PD, Jaubert P, Cole JM, Solar M, Borgquist O, Leithner C, Abed-Maillard S, Navarra L, Annborn M, Unden J, Brunetti I, Awad A, McGuigan P, Bjorkholt Olsen R, Cassina T, Vignon P, Langeland H, Lange T, Friberg H, Nielsen N; TTM2 Trial Investigators. Hypothermia versus Normothermia after Out-of-Hospital Cardiac Arrest. N Engl J Med. 2021 Jun 17;384(24):2283-2294. doi: 10.1056/NEJMoa2100591. PMID 34133859
- [Background] Zhou H, Zhu Y, Zhang Z, Lv J, Li W, Hu D, Chen X, Mei Y. Effect of arterial oxygen partial pressure inflection point on Venoarterial extracorporeal membrane oxygenation for emergency cardiac support. Scand J Trauma Resusc Emerg Med. 2021 Jul 8;29(1):90. doi: 10.1186/s13049-021-00902-5. PMID 34238331
- [Background] Kjaergaard J, Moller JE, Schmidt H, Grand J, Molstrom S, Borregaard B, Veno S, Sarkisian L, Mamaev D, Jensen LO, Nyholm B, Hofsten DE, Josiassen J, Thomsen JH, Thune JJ, Obling LER, Lindholm MG, Frydland M, Meyer MAS, Winther-Jensen M, Beske RP, Frikke-Schmidt R, Wiberg S, Boesgaard S, Madsen SA, Jorgensen VL, Hassager C. Blood-Pressure Targets in Comatose Survivors of Cardiac Arrest. N Engl J Med. 2022 Oct 20;387(16):1456-1466. doi: 10.1056/NEJMoa2208687. Epub 2022 Aug 27. PMID 36027564
- [Background] Schmidt H, Kjaergaard J, Hassager C, Molstrom S, Grand J, Borregaard B, Roelsgaard Obling LE, Veno S, Sarkisian L, Mamaev D, Jensen LO, Nyholm B, Hofsten DE, Josiassen J, Thomsen JH, Thune JJ, Lindholm MG, Stengaard Meyer MA, Winther-Jensen M, Sorensen M, Frydland M, Beske RP, Frikke-Schmidt R, Wiberg S, Boesgaard S, Lind Jorgensen V, Moller JE. Oxygen Targets in Comatose Survivors of Cardiac Arrest. N Engl J Med. 2022 Oct 20;387(16):1467-1476. doi: 10.1056/NEJMoa2208686. Epub 2022 Aug 27. PMID 36027567
- [Background] Duan J, Ma Q, Zhu C, Shi Y, Duan B. eCPR Combined With Therapeutic Hypothermia Could Improve Survival and Neurologic Outcomes for Patients With Cardiac Arrest: A Meta-Analysis. Front Cardiovasc Med. 2021 Aug 13;8:703567. doi: 10.3389/fcvm.2021.703567. eCollection 2021. PMID 34485403
- [Background] Lee JJ, Han SJ, Kim HS, Hong KS, Choi HH, Park KT, Seo JY, Lee TH, Kim HC, Kim S, Lee SH, Hwang SM, Ha SO. Out-of-hospital cardiac arrest patients treated with cardiopulmonary resuscitation using extracorporeal membrane oxygenation: focus on survival rate and neurologic outcome. Scand J Trauma Resusc Emerg Med. 2016 May 18;24:74. doi: 10.1186/s13049-016-0266-8. PMID 27193212
- [Background] Maekawa K, Tanno K, Hase M, Mori K, Asai Y. Extracorporeal cardiopulmonary resuscitation for patients with out-of-hospital cardiac arrest of cardiac origin: a propensity-matched study and predictor analysis. Crit Care Med. 2013 May;41(5):1186-96. doi: 10.1097/CCM.0b013e31827ca4c8. PMID 23388518
- [Background] Pang PYK, Wee GHL, Huang MJ, Hoo AEE, Tahir Sheriff IM, Lim SL, Tan TE, Loh YJ, Chao VTT, Soon JL, Kerk KL, Abdul Salam ZH, Sin YK, Lim CH. Therapeutic Hypothermia May Improve Neurological Outcomes in Extracorporeal Life Support for Adult Cardiac Arrest. Heart Lung Circ. 2017 Aug;26(8):817-824. doi: 10.1016/j.hlc.2016.11.022. Epub 2017 Jan 17. PMID 28159528
- [Background] Richardson ASC, Tonna JE, Nanjayya V, Nixon P, Abrams DC, Raman L, Bernard S, Finney SJ, Grunau B, Youngquist ST, McKellar SH, Shinar Z, Bartos JA, Becker LB, Yannopoulos D, B elohlavek J, Lamhaut L, Pellegrino V. Extracorporeal Cardiopulmonary Resuscitation in Adults. Interim Guideline Consensus Statement From the Extracorporeal Life Support Organization. ASAIO J. 2021 Mar 1;67(3):221-228. doi: 10.1097/MAT.0000000000001344. PMID 33627592